CLINICAL TRIAL: NCT02966964
Title: An Exploratory, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy and Safety of Tenofovir With and Without DWPUR001 in Patients With Hepatitis B Virus(HBV)
Brief Title: A Clinical Trials to Evaluate the Efficacy and Safety of Tenofovir With and Without DWPUR001 in Patients With HBV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uijeongbu St. Mary Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Chang Wook Kim, Professor, Uijeongbu St. Mary Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EURECA001
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Hepatitis; Virus, Chronic, Type B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Tenofovir 300mg qd + DWPUR001 500mg bid (Experimental): Tenofovir 300mg qd + DWPUR001 500mg bid for up to 12 months
  Interventions: Drug: DWPUR001
- Tenofovir 300mg qd + DWPUR001 300mg bid (Experimental): Tenofovir 300mg qd + DWPUR001 300mg bid for up to 12 months
  Interventions: Drug: DWPUR001
- Tenofovir 300mg qd + DWPUR001 Placebo bid (Placebo Comparator): Tenofovir 300mg qd + DWPUR001 Placebo bid for up to 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWPUR001
  Arms: Tenofovir 300mg qd + DWPUR001 300mg bid; Tenofovir 300mg qd + DWPUR001 500mg bid
Drug: Placebo
  Arms: Tenofovir 300mg qd + DWPUR001 Placebo bid

SUMMARY:
The patient who meets the inclusion/exclusion criteria is assigned to Test1 group or Test 2 group or control group randomly.

All subjects take one pill of Viread® Tab. (Tenofovir Disoproxil Fumarate 300mg) once a day for 48 weeks. At the same time, all randomized subjects take two pills of DWPUR001 or Placebo of DWPUR001 twice a day for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at the age in between 19 and 69 years at the time of agreement
2. Patients who had HBsAg-positive at least within 24 weeks or had a diagnosis with chronic hepatic disease by image test within 24 weeks from the time of screening.
3. Patients who had HBeAg-positive and HBV DNA level≥20,000 IU/mL, or HBeAg-negative and HBV DNA level≥2,000 IU/mL
4. Patients never treated with Tenofovir
5. Patients whose ALT level is more than 2 times of UNL at the time of screening
6. Patients prothrombin time prolonged≤4sec at the time of screening
7. Patients Total bilirubin level≤3.0mg/dL at the time of screening
8. Patients albumin level≥3.0g/dL at the time of screening
9. Patients ELF score≥8.5 at the time of screening
10. Patients who agree with the clinical trial voluntarily and sign on the agreement

Exclusion Criteria:

1. HIV, HCV or HDV infedted patients
2. Patients who have abnormal liver function caused by other diseases (e.g. hematochromatosis, Wilson's disease, alcoholic hepatitis, Nonalcoholic steatohepatitis, alpha 1 antitrypsin deficiency)
3. Patients who had suffered from variceal haemorrhage or hepatic encephalopathy
4. Patients who need/had liver transplant
5. Patients who have severe biliary obstruction, fulminant hepatic failure, radio-opacity gallstone, non-functional gall bladder, acute cholecystitis, Lactic acidosis/ adiposis
6. Patients who have enteritis and colitis like peptic ulcer or Crohn's disease
7. Patients who have significant kidney disease, cardiovascular disease, lung disease, nervous disease, self-immune disease, bone disease (ex: osteomalacia, osteopenia, chronic osteomyelitis, osteopsathyrosis, osteochondrosis, multiple fracture) or malignant tumor.
8. Patients who have systemic infection
9. Patients who have hypersensitivity to ursodeoxycholic acid or Tenofovir
10. Patients who have the generic problem as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
11. Patients described as below at the time of screening

    * Hb<8g/dL
    * eGFR<60mL/min/1.73m2
    * AFP level>200ng/mL or had a diagnosis with hepatocellular carcinoma based on the radiology result within 24 weeks
12. Patients who had immune- or cytokine-based antiviral agents treatment (ex. Interferon α, Peginterferon α), or immunosuppression therapy (ex. Cyclosporine, Tacrolimus) in 24 weeks at the time of screening
13. Patients who have to use the contraindication of comedication drugs during clinical trial or can't get the wash-out period
14. Women of child-bearing potential not using an effective birth control method
15. Patients who have psychiatric disorders or drug or alcohol abuse, so can't understand the purpose and process of this clinical trial
16. Patients who participated in other clinical trial in 30 days prior to the enrollment in this study
17. Patients who were determined inappropriate by the investigator to participate in this study

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of normalization of ALT level (≤1× ULN)(%) | At the 4 weeks

SECONDARY OUTCOMES:
The proportion of normalization of ALT level (≤1× ULN)(%) | At the 2, 8, 12, 24, 36, 48 weeks
The change of fibrosis marker(ELF score) compared with the baseline | At the 48 weeks
The change of immunological marker(PD-1, CTLA-4, FoxP3) compared with baseline | At the 12, 24, 48 weeks
The change of anti-oxidant/anti-inflammatory marker(SOD, MDA, TNF-α) | At the 24, 48 weeks
The change of HBV DNA level compared with baseline (IU/mL) | At the 12, 24, 36, 48 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Korea University Ansan Hospital, Ansan-si
  - Bundang CHA medical center, Bundang
  - Incheon St. Mary Hospital, Incheon
  - Severance Hospital, Seoul
  - Ajou University Medical Center, Suwon
  - Uijeongbu St. Mary Hospital, Uijongbu